CLINICAL TRIAL: NCT01185860
Title: A Multiple-Dose Study To Evaluate Safety, Tolerability, Pharmacokinetics and Antiviral Activity of Ritonavir-Boosted RO5190591 in Combination With Peginterferon Alfa-2a Plus Ribavirin in Patients With Chronic Hepatitis C Genotype 1
Brief Title: A Study of Ritonavir-Boosted Danoprevir (RO5190591) in Combination With Pegasys and Ribavirin in Patients With Chronic Hepatitis C Genotype 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NP22660; 2009-012426-36
Record Dates: First submitted 2010-08-19; First posted 2010-08-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — danoprevir; peginterferon alfa-2a; Ribavirin; Ritonavir

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- A (Active Comparator)
  Interventions: Drug: danoprevir; Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin
- B (Experimental)
  Interventions: Drug: danoprevir; Drug: peginterferon alfa-2a [Pegasys]; Drug: ribavirin; Drug: ritonavir
- C (Placebo Comparator)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]; Drug: placebo; Drug: ribavirin; Drug: ritonavir

INTERVENTIONS:
Drug: danoprevir — oral doses
  Arms: A; B
Drug: peginterferon alfa-2a [Pegasys] — 180 mcg sc once weekly
Drug: placebo — oral doses
  Arms: C
Drug: ribavirin — 1000-1200mg/day po
Drug: ritonavir — oral doses
  Arms: B; C

SUMMARY:
This study will evaluate the efficacy, safety and tolerability of danoprevir (RO5190591) plus ritonavir as compared to danoprevir alone or placebo plus ritonavir in patients with chronic hepatitis C genotype 1 receiving Pegasys (peginterferon alfa-2a) and ribavirin. Patients in cohorts will be randomized to receive either oral doses of danoprevir, or danoprevir plus ritonavir, or placebo plus ritonavir. All patients will receive Pegasys (180mcg sc once weekly) plus ribavirin (1000-1200mg/day po), with the option to continue this treatment after completion of study drug treatment. Anticipated time on study treatment is up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18-65 years of age
* Chronic hepatitis C genotype 1
* HCV treatment naïve, or without sustained virologic response on prior PEG-INF/RBV treatment
* Body mass index (BMI) 18 - 35 kg/m2, inclusive; minimum weight 45 kg

Exclusion Criteria:

* Liver cirrhosis
* Decompensated liver disease or impaired liver function
* Medical condition associated with chronic liver disease other than chronic hepatitis C
* Positive for hepatitis B or HIV infection at screening
* History of alcohol consumption exceeding 2 standard drinks per day when averaged over the course of a given week

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Adverse events, ECG, laboratory parameters | approximately 3 years
Pharmacokinetics: Cmax, AUC, Cmin, Tmax, Cl, T1/2 | Days 3-9
Antiviral activity: HCV RNA (COBAS Taqman HCV Test) | from baseline to Day 28

SECONDARY OUTCOMES:
Viral resistance development | from baseline to Day 17
Effects on cytochrome P450(CYP)2C9 and 3A isozymes | from baseline to Day 17
Virological response in prior null-responders | from baseline to week 72
Comparison of pharmacokinetics and antiviral activity between treatment-naïve patients and prior null-responders to standard of care treatment | approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Montpellier, France
- New Zealand (2):
  - Christchurch
  - Grafton
- Warsaw, Poland

REFERENCES:
- [Derived] Gane EJ, Rouzier R, Wiercinska-Drapalo A, Larrey DG, Morcos PN, Brennan BJ, Le Pogam S, Najera I, Petric R, Tran JQ, Kulkarni R, Zhang Y, Smith P, Yetzer ES, Shulman NS. Efficacy and safety of danoprevir-ritonavir plus peginterferon alfa-2a-ribavirin in hepatitis C virus genotype 1 prior null responders. Antimicrob Agents Chemother. 2014;58(2):1136-45. doi: 10.1128/AAC.01515-13. Epub 2013 Dec 2. PMID 24295986
- [Derived] Morcos PN, Chang L, Kulkarni R, Giraudon M, Shulman N, Brennan BJ, Smith PF, Tran JQ. A randomised study of the effect of danoprevir/ritonavir or ritonavir on substrates of cytochrome P450 (CYP) 3A and 2C9 in chronic hepatitis C patients using a drug cocktail. Eur J Clin Pharmacol. 2013 Nov;69(11):1939-49. doi: 10.1007/s00228-013-1556-y. Epub 2013 Jul 20. PMID 23872824
- [Derived] Gane EJ, Rouzier R, Stedman C, Wiercinska-Drapalo A, Horban A, Chang L, Zhang Y, Sampeur P, Najera I, Smith P, Shulman NS, Tran JQ. Antiviral activity, safety, and pharmacokinetics of danoprevir/ritonavir plus PEG-IFN alpha-2a/RBV in hepatitis C patients. J Hepatol. 2011 Nov;55(5):972-9. doi: 10.1016/j.jhep.2011.01.046. Epub 2011 Feb 24. PMID 21354234